CLINICAL TRIAL: NCT07238023
Title: Testing the Feasibility and Acceptability of a Remotely Delivered Program to Promote Active Living Among People With Metastatic Breast Cancer
Brief Title: Promoting Active Living Among People With Metastatic Breast Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: TSET Health Promotion Research Center (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 18941
Record Dates: First submitted 2025-09-29; First posted 2025-11-20 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Invasive Breast Cancer
Keywords: aerobic physical activity; muscle strengthening physical activity; mindfulness; acceptance; telehealth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acceptance- and Mindfulness-Based Intervention (Experimental): Provision of standard self-regulatory behavior change techniques, plus acceptance and mindfulness-based physical activity promotion
  Interventions: Behavioral: Acceptance- and mindfulness-based physical activity promotion

INTERVENTIONS:
Behavioral: Acceptance- and mindfulness-based physical activity promotion — This intervention will be delivered over the course of up to 8-12 weeks.
  It will include:
  1. the provision of a wearable physical activity tracker
  2. empirically supported behavior change techniques for promoting physical activity
  3. Acceptance and Commitment Therapy-informed didactic content centered on promoting physical activity
  4. a social component with game design elements reflecting acceptance and mindfulness practices (i.e., the ability to share responses to "Weekly Challenges" and view and comment on others' entries).

SUMMARY:
Individuals with metastatic breast cancer are living longer but often face persistent fatigue, functional decline, and psychological distress. Physical activity is generally safe for this population and may alleviate symptom burden. Yet, limited interventions are tailored to the unique and needs and preferences of this population. This study aims to evaluate the acceptability and feasibility of a mindfulness- and acceptance-based physical activity program designed to support mental, social, and spiritual well-being among people with metastatic breast cancer. A single group, pretest-posttest trial (N=38) will be conducted to inform scalable strategies to promote active living and enhance quality of life among people with advanced cancer.

ELIGIBILITY:
Inclusion Criteria:

* having been diagnosed with metastatic breast cancer
* medical clearance from healthcare provider to participate in this study
* life expectancy of at least 6 months as per the participant's healthcare provider
* Eastern Cooperative Oncology Group performance status of or 0 or 1
* being willing and able to use a smartphone and web interface with or without assistance; if assistance is needed, it must be readily available
* adequate visual and hearing acuity to use a smartphone and web interface as indicated by self-report
* adequate motor capacity to use a smartphone and web interface as indicated by self-report
* willingness to download and use study-specific app(s), the Fitbit mobile application (this requires use of a Google Gmail account), and other mobile applications for study purposes as needed
* completed baseline survey

Exclusion Criteria:

* contraindications to physical activity (e.g., uncontrolled hypertension or cardiac disease noted by the patient's treating healthcare provider)
* presence of bone metastases deemed unstable by the treating healthcare provider.
* untreated brain metastases
* history of dementia or other major neurocognitive disorder
* received a diagnosed of Major Depressive Disorder within the previous 6 months
* received a diagnosis of a major psychiatric conditions such as bipolar disorder, psychosis, schizophrenia, or alcoholism that could affect the ability to understand and/or complete the study
* currently hospitalized
* enrolled in hospice
* inability to speak, read, and write in English at the 7th grade level

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Semi-structured Interviews | Week 9
  Semi-structured interviews will be used to assess participants' overall experience and their perceptions of the usability, usefulness, and enjoyability of the intervention.
Perceived ease of use | Week 9
  Face valid questions will be used to determine whether participants found the interventions easy to use. The face valid questions consists of five 7-point Likert-type items. Responses range from "Not At All Easy" (scored as 1) to "Very Easy" (scored as 7). Higher scores reflect greater ease of use.
Perceived Usefulness | Week 9
  Face valid questions will be used to determine whether participants found the interventions useful. The face valid questions consists of five 7-point Likert-type items. Responses range from "Not At All Useful" (scored as 1) to "Very Useful" (scored as 7). Higher scores reflect greater perceived usefulness.
Enjoyability - Face Valid Questions | Week 9
  Face valid questions will be used to assess the enjoyability of the interventions in this study. The face valid questions consists of five 7-point Likert-type items. Responses range from "Not At All Enjoyable" (scored as 1) to "Very Enjoyable" (scored as 7). Higher scores reflect greater enjoyability.
Enjoyability - Interest/Enjoyment Subscale | Week 9
  The interest/enjoyment subscale of the Intrinsic Motivation Inventory (IMIe) will be used to assess the enjoyability of the interventions in this study. The IMIe sub-scale consists of seven 7-point Likert-type items. Responses range from "Not At All True" (scored as 1) to "Very True" (scored as 7). Higher scores reflect greater enjoyability.
Feasibility of the Program - Study Retention | Week 9
  We will assess program feasibility via measurements of study retention. We will compute what percentage of enrolled participant complete post-intervention data collection procedures.
Feasibility of the Program - Adherence | Week 9
  We will assess program feasibility via measurements of intervention adherence. We will compute what percentage of participants engage with at least 75% of the intervention modules.
Feasibility of Collecting Biological Samples | Week 9
  We will assess the feasibility of assessing gene expression in the present context by assessing what percentage of enrolled participants provide analyzable data in optional post-intervention blood draws.

OTHER OUTCOMES:
Physical Activity | Baseline; Week 9
  A modified Godin Leisure-Time Exercise Questionnaire will be used to assess participants' physical activity patterns. This self-report measure assesses the number of minutes of strenuous-, moderate-, and light-intensity exercise in a typical week. An additional item will be included that assesses the number of bouts of muscle-strengthening exercise in a typical week. We will also gather data provided by consumer-grade, wearable physical activity trackers (Fitbit Charge series or similar).
Feelings of Vitality | Baseline; Week 9
  The Subjective Vitality Scale (SVS) will be used to will be used to assess participants' feelings of vitality. The SVS consists of seven 7-point Likert-type items. Responses range from "Not At All True" (scored as 1) to "Very True" (scored as 7). Higher scores reflect greater enjoyability.
Meaning Salience | Baseline; Week 9
  The Meaning Awareness Scale (MAS) will be used to assess meaning salience. The MAS consists of six 7-point Likert-type items. Responses range from "Very Rarely" (scored as 1) to "Very Often" (scored as 7). Higher scores reflect greater meaning salience.
Psychological Flexibility | Baseline; Week 9
  The Personalized Psychological Flexibility Index (PPFI) will be used to assess psychological flexibility. The PPFI consists of sixteen 7-point Likert-type items. Responses range from "Strongly Disagree" (scored as 1) to "Strongly Agree" (scored as 7). Higher scores reflect greater psychological flexibility.
Physical Activity Motivation | Baseline; Week 9
  The Behavioral Regulation for Exercise Questionnaire-4 (BREQ-4) will be used to assess physical activity motivation. The BREQ-4 consists of twenty-eight 5-point Likert-type items. Responses range from "Not True For Me" (scored as 0) to "Very True For Me" (scored as 4). It is best practice to score each of the seven subscales separately (i.e., obtain separate scores for amotivation, external regulation, introjected avoidance regulation, introjected approach regulation, identified regulation, integrated regulation, and intrinsic regulation). For each subscale, higher scores reflect greater usage of that type of regulation.
Physical Activity Acceptance | Baseline; Week 9
  The Physical Activity Acceptance Questionnaire (PAAQ) will be used to assess physical activity acceptance. The PAAQ consists of ten 7-point Likert-type items. Responses range from "Never True" (scored as 1) to "Always True" (scored as 7). It is best practice to score each of the two subscales separately (i.e., obtain separate scores for cognitive acceptance and behavioral commitment). For each subscale, higher scores reflect greater acceptance/commitment.
Health-Related Quality of Life - Physical Function | Baseline; Week 9
  The Patient-Reported Outcomes Measurement Information System-29 (PROMIS-29+2 Profile v2.1) will be used to assess health-related quality of life. The PROMIS-29+2 Profile v2.1 consists of thirty-one items spanning nine subscales (i.e., physical function, anxiety, depressive symptoms, fatigue, sleep disturbance, ability to participate in social roles and activities, pain interference, cognition, and pain intensity). The physical function subscale has 4 items with 5-point Likert-type responses (e.g., ranging from "Unable To Do" (scored as 1) to "Without Any Difficulty" (scored as 5). Higher scores for physical function are favorable.
Health-Related Quality of Life - Anxiety | Baseline; Week 9
  The Patient-Reported Outcomes Measurement Information System-29 (PROMIS-29+2 Profile v2.1) will be used to assess health-related quality of life. The PROMIS-29+2 Profile v2.1 consists of thirty-one items spanning nine subscales (i.e., physical function, anxiety, depressive symptoms, fatigue, sleep disturbance, ability to participate in social roles and activities, pain interference, cognition, and pain intensity). The anxiety subscale has 4 items with 5-point Likert-type responses (e.g., ranging from "Never" (scored as 1) to "Always" (scored as 5). Higher scores for anxiety are not favorable.
Health-Related Quality of Life - Depressive Symptoms | Baseline; Week 9
  The Patient-Reported Outcomes Measurement Information System-29 (PROMIS-29+2 Profile v2.1) will be used to assess health-related quality of life. The PROMIS-29+2 Profile v2.1 consists of thirty-one items spanning nine subscales (i.e., physical function, anxiety, depressive symptoms, fatigue, sleep disturbance, ability to participate in social roles and activities, pain interference, cognition, and pain intensity). The depressive symptoms subscale has 4 items with 5-point Likert-type responses (e.g., ranging from "Never" (scored as 1) to "Always" (scored as 5). Higher scores for depressive symptoms are not favorable.
Health-Related Quality of Life - Fatigue | Baseline; Week 9
  The Patient-Reported Outcomes Measurement Information System-29 (PROMIS-29+2 Profile v2.1) will be used to assess health-related quality of life. The PROMIS-29+2 Profile v2.1 consists of thirty-one items spanning nine subscales (i.e., physical function, anxiety, depressive symptoms, fatigue, sleep disturbance, ability to participate in social roles and activities, pain interference, cognition, and pain intensity). The fatigue subscale has 4 items with 5-point Likert-type responses (e.g., ranging from "Not At All" (scored as 1) to "Very Much" (scored as 5). Higher scores for fatigue are not favorable.
Health-Related Quality of Life - Sleep Disturbance | Baseline; Week 9
  The Patient-Reported Outcomes Measurement Information System-29 (PROMIS-29+2 Profile v2.1) will be used to assess health-related quality of life. The PROMIS-29+2 Profile v2.1 consists of thirty-one items spanning nine subscales (i.e., physical function, anxiety, depressive symptoms, fatigue, sleep disturbance, ability to participate in social roles and activities, pain interference, cognition, and pain intensity). The sleep disturbance subscale has 4 items with 5 point Likert-type responses (e.g., ranging from "Not At All" (scored as 1) to "Very Much" (scored as 5). Higher scores indicate more sleep disturbance.
Health-Related Quality of Life - Ability to Participate in Social Roles and Activities | Baseline; Week 9
  The Patient-Reported Outcomes Measurement Information System-29 (PROMIS-29+2 Profile v2.1) will be used to assess health-related quality of life. The PROMIS-29+2 Profile v2.1 consists of thirty-one items spanning nine subscales (i.e., physical function, anxiety, depressive symptoms, fatigue, sleep disturbance, ability to participate in social roles and activities, pain interference, cognition, and pain intensity). The ability to participate in social roles and activities subscale has 4 items with 5 point Likert-type responses (e.g., ranging from "Not At All" (scored as 1) to "Very Much" (scored as 5). Higher scores for ability to participate in social roles and activities are not favorable.
Health-Related Quality of Life - Pain Interference | Baseline; Week 9
  The Patient-Reported Outcomes Measurement Information System-29 (PROMIS-29+2 Profile v2.1) will be used to assess health-related quality of life. The PROMIS-29+2 Profile v2.1 consists of thirty-one items spanning nine subscales (i.e., physical function, anxiety, depressive symptoms, fatigue, sleep disturbance, ability to participate in social roles and activities, pain interference, cognition, and pain intensity). The pain interference subscale has 4 items with 5 point Likert-type responses (e.g., ranging from "Not At All" (scored as 1) to "Very Much" (scored as 5). Higher scores for pain interference are not favorable.
Health-Related Quality of Life - Cognition | Baseline; Week 9
  The Patient-Reported Outcomes Measurement Information System-29 (PROMIS-29+2 Profile v2.1) will be used to assess health-related quality of life. The PROMIS-29+2 Profile v2.1 consists of thirty-one items spanning nine subscales (i.e., physical function, anxiety, depressive symptoms, fatigue, sleep disturbance, ability to participate in social roles and activities, pain interference, cognition, and pain intensity). The cognition subscale has 2 items with 5-point Likert-type responses (e.g., ranging from "Not At All" (scored as 1) to "Very Much" (scored as 5). Higher scores for cognition are favorable.
Health-Related Quality of Life - Pain Intensity | Baseline; Week 9
  The Patient-Reported Outcomes Measurement Information System-29 (PROMIS-29+2 Profile v2.1) will be used to assess health-related quality of life. The PROMIS-29+2 Profile v2.1 consists of thirty-one items spanning nine subscales (i.e., physical function, anxiety, depressive symptoms, fatigue, sleep disturbance, ability to participate in social roles and activities, pain interference, cognition, and pain intensity). The pain intensity subscale has 1 item with responses ranging from "No Pain" (scored as 0) to "Worst Pain Imaginable" (scored as 10). Higher scores for pain intensity are not favorable.

IPD SHARING:
Plan to Share IPD: Undecided
We are undecided about sharing individual participant data at this time. This study involves a sensitive population and may result in a relatively small sample size, which increases the risk of participant re-identification even after de-identification procedures. We will evaluate data sharing feasibility after study completion, taking into account participant privacy protections, ethical considerations, and institutional policies.